CLINICAL TRIAL: NCT04915456
Title: Prospective Randomized, Placebo-controlled Clinical Study to Study the Effect of Postoperative Additive Systemic Steroids in Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Effect of Postoperative Additive Systemic Steroids in CRSwNP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Sarina Mueller, PD Dr. med., Friedrich-Alexander-Universität Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP1
Record Dates: First submitted 2021-05-24; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Sinusitis, Chronic
Keywords: steroid; recurrence; smell; biomarker; endoscopy
MeSH Terms: conditions — Sinusitis; Bronchiolitis Obliterans Syndrome; Recurrence; Anosmia | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic steroid (Prednisolone) (Experimental): Prednisolone 50mg (tapered down until postoperative day (POD) 14, then 5mg for 14 days), tablets
  Interventions: Drug: Systemic Steroid (Prednisolone)
- Placebo (Placebo Comparator): Lactose monohydrate, tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Systemic Steroid (Prednisolone) — Systemic steroids (Prednisolone) additive to topical steroids (Mometasone fuorate) in a postoperative setting after FESS
  Arms: Systemic steroid (Prednisolone)
Other: Placebo — Placebo additive to topical steroids in a postoperative setting after FESS
  Arms: Placebo

SUMMARY:
This study investigate the additive effect of systemic postoperative steroids in patients with chronic rhinosinusitis (CRSwNP). All patients receive a functional endoscopic sinus surgery (FESS) followed by topical steroid spray for 3 months. Postoperatively, patients will be randomized to either an additional systemic steroid or a placebo for 1 month. Patients will be followed for 2 years. Effect on Nasal Polyp score (NPS), Lund-Kennedy-Score (LKS), recurrence rates, smell scores, Rhinosinusitis Disability Index (RSDI), Short-Form 36 (SF-36) and mucus/serum biomarkers will be measured.

ELIGIBILITY:
Inclusion Criteria:

* CRSwNP
* refractory to medical therapy
* no previous sinus surgery
* Lund-Kennedy-Score ≥ 1
* Lund-Mackay-Score ≥ 10

Exclusion Criteria:

* ciliary impairment
* autoimmune disease
* cystic fibrosis
* immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-01-18 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Nasal Polyp Score (NPS) | first visit until 24 months, change is measured between baseline and each follow-up time point up to 24 months (follow-up time points are as follows: 3 weeks, 3 months, 6 months, 9 months, 12 months, 18 months)
  Each nostril will be assessed separately. The highest score will be graded. Each nostril will be scored from 0-4 (0=no polyps, 1=polyps confined to the middle meatus, 3=polyps extending beyond middle meatus, 4=large polyps causing almost complete nasal obstruction)

SECONDARY OUTCOMES:
Lund-Kennedy-Score (LKS) | first visit until 24 months, change is measured between baseline and each follow-up time point up to 24 months (follow-up time points are as follows: 3 weeks, 3 months, 6 months, 9 months, 12 months, 18 months)
  Lund-Kennedy-Scores range from 0-12. Scoring includes the assessment of polyps (0=no polyps, 1=middle meatus, 2= beyond middle meatus), discharge (0=no discharge, 1=thin discharge, 2=edema/scarring/crusting (0=absent, 1=mild, 2=severe)
Smell Scores | first visit until 24 months, change is measured between baseline and each follow-up time point up to 24 months (follow-up time points are as follows: 3 weeks, 3 months, 6 months, 9 months, 12 months, 18 months)
  Sniffing Sticks Screening-16 test ("forced choice"), graded from 0-16 with a higher score indicating a better sense of smell, anosmia is defined as a score ≤7
Recurrence rates | first visit until 24 months, change is measured between baseline and each follow-up time point up to 24 months (follow-up time points are as follows: 3 weeks, 3 months, 6 months, 9 months, 12 months, 18 months)
  Increase of NPS per side ≥ 2 within 2 year follow-up
Sinonasal Symptom Score | first visit until 24 months, change is measured between baseline and each follow-up time point up to 24 months (follow-up time points are as follows: 3 weeks, 3 months, 6 months, 9 months, 12 months, 18 months)
  nasal congestion, anterior rhinorrhea, posterior rhinorrhea, sneezing, pruritus in the nose, tearing, ear pressure, throat pain, facial pain or pressure, headache, numbness in cheek/lips/teeth. All graded from 0-3 (0=no problems, 1=mild problems, 2= moderate problems, 3= severe problems)
Mucus and serum biomarker levels | first visit until 24 months, change is measured between baseline and each follow-up time point up to 24 months (follow-up time points are as follows: 3 weeks, 3 months, 6 months, 9 months, 12 months, 18 months)
  Pappalysin-1, Cystatin-SN, Periostin, SerpinE1, SerpinF2 (measured in pg/ml)
RSDI (Rhinosinusitis Disability Index) | first visit until 24 months, change is measured between baseline and each follow-up time point up to 24 months (follow-up time points are as follows: 3 weeks, 3 months, 6 months, 9 months, 12 months, 18 months)
  validated 30-item Likert scale instrument containing three subscales that assess the impact of sinusitis on physical, functional, and emotional domains. The Score ranges from 0-120. Higher total and subscale RSDI scores represent a worse impact of sinus disease.
SF-36 (Short Form-36) | first visit until 24 months, change is measured between baseline and each follow-up time point up to 24 months (follow-up time points are as follows: 3 weeks, 3 months, 6 months, 9 months, 12 months, 18 months)
  There is no single overall score for the SF-36, instead, it generates 8 subscales and two summary scores. The subscales are: physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role-limitations due to emotional problems, mental health. The scoring ranges from 0-100. Higher total and subscale scores represent a better health situation.